CLINICAL TRIAL: NCT06982846
Title: A Randomized, Placebo-Controlled, Parallel Study to Investigate the Response of Participants With Type 2 Diabetes Mellitus on Once-Weekly Retatrutide to Hypoglycemia
Brief Title: A Study to Investigate the Response of Participants With Type 2 Diabetes Mellitus on Once-Weekly Retatrutide to Hypoglycemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27316; J1I-MC-GZQF (Other: Eli Lilly and Company); 2024-518471-63-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retatrutide (Experimental): Participants will receive escalated doses of retatrutide administered subcutaneously (SC) every week (QW) until reaching target dose.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive matching placebo administered SC QW.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the effect of retatrutide versus placebo, administered every week, on time to recovery from hypoglycemia during hypoglycemic clamp in participants with Type 2 Diabetes Mellitus (T2DM) following 16 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with T2DM for at least 6 months prior to screening.
* Treated with diet and exercise and stable treatment with metformin with or without 1 additional allowed oral antihyperglycemic medications (OAM), 3 months prior to screening.

  * Treatment with metformin will be considered stable if all prescribed total daily doses for this period were ±850 mg from the original prescription for the same participant.
  * Allowed OAMs include dipeptidyl peptidase-4 (DPP-IV) inhibitors, sodium-glucose co-transporter-2 (SGLT2) inhibitors, glinides, or sulfonylureas.
* Have a hemoglobin A1c value at screening of

  * ≥6.0% (≥ 42 millimole per liter(mmol/L)) and ≤9.5% (≤80 mmol/L) if on metformin only or
  * ≥6.0% (≥42 mmol/L) and ≤8.5% (≤69 mmol/L) if on metformin in combination with 1 additional allowed OAM.
* Have a BMI within the range 25.0 kg/m2 and 45.0 kg/m2 kg/m2 (both inclusive).
* Have had a stable body weight that is less than 5% change in body weight for more than 3 months prior to screening.

Exclusion Criteria:

* Have Type 1 diabetes mellitus.
* Have had more than 1 episode of severe hypoglycemia, as defined by the American Diabetes Association criteria, within 6 months before screening or has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms.
* Have had 1 or more episodes of ketoacidosis or hyperosmolar state/coma requiring hospitalization within the 6 months prior to screening.
* Have impaired renal estimated glomerular filtration rate <60 mL/min/1.73 m2 calculated by Chronic Kidney Disease-Epidemiology.
* Have acute or chronic pancreatitis or a history of acute idiopathic pancreatitis.
* Have elevations in

  * serum aspartate aminotransferase (AST) >2.5× upper limit normal (ULN)
  * serum alanine aminotransferase (ALT) >2.5×ULN
  * total bilirubin level (TBL) >1.5×ULN, or
  * alkaline phosphatase (ALP) level ≥1.5× ULN.
* Have a known clinically significant gastric emptying abnormality.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time-to-Event of Recovery of Plasma Glucose (PG) Concentration from 48 Milligram per Deciliter (48 mg/dL) to 70 mg/dL (tPG_nadir-70 mg/dL) | Within 60 minutes after nadir
  Time-to-event of recovery of PG concentration from 48 mg/dL to 70 mg/dL.

SECONDARY OUTCOMES:
Time to Reach Recovery of Plasma Glucose (PG) Concentration from 48 mg/dL to 70 mg/dL (tPG_nadir-70 mg/dL) Including Recovery Beyond 60 Minutes. | Beyond 60 minutes after nadir
  Time-to-event of recovery of PG concentration from 48 mg/dL to 70 mg/dL including recovery beyond 60 minutes.
Percentage of Participants Who Require Rescue Glucose Infusion to Attain Recovery PG Concentration of 70 mg/dL | Up to 60 minutes after nadir
  Percentage of participants who require rescue glucose infusion to attain recovery PG concentration of 70 mg/dL.
Hypoglycemic Symptoms Score at set PG Concentration Points | Day 114 during hypoglycemic clamp
  Hypoglycemia symptoms were measured with the Edinburgh Hypoglycemia Symptom Scale (EHSS) where lower scores indicate fewer symptoms.
Percentage of Participants Who Experienced Hypoglycemic Awareness at Set PG Points | Day 114 during hypoglycemic clamp
  Percentage of participants who experienced hypoglycemic awareness at set PG points.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Medizinische Universität Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No